CLINICAL TRIAL: NCT05232760
Title: SUPER-DIALYSIS-Study: Supera Stent Interventions in Juxta-anastomotic (re)Stenosis
Status: Completed | Type: Observational
Sponsor: Klinikum Arnsberg (Other)
Responsible Party: Sponsor
Other Study IDs: ASL202002
Record Dates: First submitted 2021-11-23; First posted 2022-02-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Stenosis of Arteriovenous Dialysis Fistula
Keywords: Juxta-anastomotic stenose of arteriovenous fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SUPERA peripheral stent system
  Interventions: Device: Supera™ Peripheral Stent System

INTERVENTIONS:
Device: Supera™ Peripheral Stent System — The device will be employed for treatment of juxta-anastomotic stenosis in failing AV fistula after previous percutaneous angioplasty procedures

SUMMARY:
The purpose of this exploratory study is to evaluate safety and effectiveness of treatment of juxta-anastomotic (re)stenosis with SUPERA stent by improving hemodynamic situation through obtuse shaping of the anastomosis.

DETAILED DESCRIPTION:
Up to 50 patients undergoing percutaneous intervention due to juxta-anastomotic (re-)stenosis of the AV fistulas will be enrolled in this single-arm, prospective, multi-center CE marked study (IIT). Hemodialysis patients with failing radial-cephalic arteriovenous fistula (AVF) will receive treatment with the SUPERA stent and will be followed-up at 1, 3, 6 and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years of age, able to perform follow-up visits, have a life expectancy > 12 months.
2. Hemodialysis patients undergoing endovascular angioplasty due to a clinically symptomatic stenosis (de novo or restenosis) of the juxta-anastomotic radiocephalic AVF with significant stenosis (lumen diameter < 2.7mm)
3. Patients with at least one previous endovascular intervention to restore AVF function
4. The target lesion consists of one or more lesions with a target lesion length of less than or equal to 80 mm in the juxta-anastomotic segment of the radiocephalic AVF
5. The target blood vessel diameter of the target lesion is between 4.0 and 7.5 mm (in angiographic or ultrasound evaluation)
6. If there are other non-target lesions, then non-target lesions must be successfully cured with a balloon before treating the target lesion

Exclusion Criteria:

1. Patients with AVF stenosis observed and estimated as nonsignificant (lumen diameter > 2.7mm) or a vessel <4.0 and > 7.5 mm in diameter by visual estimation
2. Patients with a known hypersensitivity or contraindication to anticoagulant/anti-platelet therapies, or sensitivity to contrast media that cannot be adequately pre-medicated.
3. Patients with any contraindications as mentioned in the Instructions for Use (IFU) of the study device.
4. Patients that are currently participating in another clinical trial involving any investigational drug or device that may potentially confound the results of the study, or that would limit the patient's compliance with the follow-up requirements of the study.
5. Prior enrolment in this trial
6. Women who are pregnant or lactating
7. Patients, who underwent a major surgery (such as thoracotomy, craniotomy, etc.) within 30 days prior to the study.
8. Patients, who have scheduled a major surgery (such as thoracotomy, craniotomy, etc.). within 30 days after enrolment -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients from clinics with vascular centers
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with primary patency of juxta-anastomose at month 3 | 3 months
  Primary patency is defined as clinically assessed intervention free (IFP) period

SECONDARY OUTCOMES:
Number of patients with primary patency of juxta-anastomose | 1, 6 and 12 months.
  Primary patency is defined as clinically assessed intervention free (IFP) period
Number of patients with assisted primary patency | 1, 3, 6 and 12 months
  Assisted primary patency is defined as interval until access thrombosis or the time of measurement of patency, including intervening manipulations (surgical or endovascular interventions) designed to maintain the functionality of a patent access
Number of patients with secondary patency | 1, 3, 6 and 12 months
  Secondary patency is defined as interval until access abandonment, thrombosis, or the time of patency measurement including intervening manipulations (surgical or endovascular interventions) designed to reestablish functionality in thrombosed access
Number of patients with technical success | Day 1 after the index procedure
  Residual stenosis < 30% after treatment with Supera stent (measured by angiography during the procedure)
Number of patients with procedural success | 1 day (discharge)
  Residual stenosis < 30% with no major adverse events (MAE)
Number of patients with clinical success | 1 day (discharge)
  Hemodialysis access function improved, dialysis function restored, and at least one dialysis session completed after the procedure until discharge
Number of patients with access circuit patency | 1,3,6,12 months
  Freedom from development of a stenosis in any region of the AVF circuit, including the juxta-anastomotic segment
Recirculation rate | 1, 3, 6 and 12 months
Fistula flow | 1, 3, 6 and 12 months
  Flow in AV fistula measured with ultrasound
Incidence of major adverse events | 6 and 12 months
  Major adverse events (death, stroke)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lichtenberg, Dr.med., Principal Investigator — Klinikum Hochsauerland GmbH
Locations (1):
- Klinikum Hochsauerland GmbH, Arnsberg, Germany